CLINICAL TRIAL: NCT07224100
Title: Phase II Study of Dose-Adjusted EPOCH ± Rituximab + Ponatinib for Adults With Newly-Diagnosed Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: Dose-Adjusted EPOCH With or Without Rituximab Plus Ponatinib for the Treatment of Newly-Diagnosed Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia/Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125799; NCI-2025-07631 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-10-29; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; B Lymphoblastic Leukemia/Lymphoma With t(9;22)(q34.1;q11.2); BCR-ABL1; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; pegylated granulocyte colony-stimulating factor; ponatinib; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (DA-EPOCH, rituximab, ponatinib) (Experimental): Patients receive etoposide IV, doxorubicin IV, and vincristine IV over 96 hours on days 1-4, cyclophosphamide IV over 1 hour on day 5, and prednisone PO BID on days 1-5 and ponatinib PO QD on days 1-21 of each cycle. Patients receive filgrastim SC on day 6, 7, or 8 and continue until ANC > 2000/µL past nadir or pegfilgrastim SC on day 6, 7, or 8 of each cycle. Patients who are CD20 positive also receive rituximab IV on day 1 or 5 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, bone marrow aspiration and biopsy and CT throughout the study. Additionally, patients may undergo PET/CT at enrollment.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Biological: Filgrastim; Biological: Pegfilgrastim; Drug: Ponatinib; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
Drug: Ponatinib — Given PO
  Other Names: AP 24534; AP-24534; AP24534
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Computed Tomography — Undergo CT and PET/CT
  Other Names: CAT; CAT scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography (CT) scan; CT; CT scan; Diagnostic CAT Scan
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET scan; Positron Emission Tomography Scan; PT

SUMMARY:
This phase II trial tests the effect of dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (DA-EPOCH) with or without rituximab plus ponatinib in treating patients newly diagnosed with Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia or lymphoma (ALL). Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and deoxyribonucleic acid (DNA) repair and may kill cancer cells. Prednisone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Vincristine is in a class of medications called vinca alkaloids. It works by stopping cancer cells from growing and dividing and may kill them. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells. It may also lower the body's immune response. Doxorubicin is a drug that is used to treat many types of cancer and is being studied in the treatment of other types of cancer. Doxorubicin comes from the bacterium Streptomyces peucetius. It damages DNA and may kill cancer cells. It is a type of anthracycline antitumor antibiotic. DA-EPOCH involves a longer exposure time to doxorubicin, vincristine and etoposide compared to a higher concentration over a shorter time which may provide better tumor response. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Ponatinib blocks BCR::ABL1 and other proteins, which may help keep cancer cells from growing and may kill them. It may also prevent the growth of new blood vessels that tumors need to grow. Ponatinib is a type of tyrosine kinase inhibitor and a type of antiangiogenesis agent. Giving DA-EPOCH with or without rituximab plus ponatinib may be safe, tolerable, and/or effective in treating patients with newly diagnosed Ph+ ALL.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive etoposide intravenously (IV), doxorubicin IV, and vincristine IV over 96 hours on days 1-4, cyclophosphamide IV over 1 hour on day 5, and prednisone orally (PO) twice daily (BID) on days 1-5 and ponatinib PO once daily (QD) on days 1-21 of each cycle. Patients receive filgrastim subcutaneously (SC) on day 6, 7, or 8 and continue until absolute neutrophil count (ANC) > 2000/µL past nadir or pegfilgrastim SC on day 6, 7, or 8 of each cycle. Patients who are CD20 positive also receive rituximab IV on day 1 or 5 of each cycle. Cycles repeat every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, bone marrow aspiration and biopsy and computed tomography (CT) throughout the study. Additionally, patients may undergo positron emission tomography (PET)/CT at enrollment.

After completion of study treatment, patients are followed every 3 months for 2 years, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and older) with newly-diagnosed Ph+ B-ALL. Ph status will be determined by routine cytogenetics, fluorescence in situ hybridization (FISH), and/or reverse transcriptase-polymerase chain reaction (RT-PCR) for the BCR::ABL1 translocation
* Marrow or blood involvement by abnormal lymphoblasts detectable by multiparameter flow cytometry (MFC)
* Total bilirubin (TBili) ≤ 1.5 x upper limit of normal (ULN) (unless attributed to Gilbert's disease or other causes of inherited indirect hyperbilirubinemia, at which point TBili must be ≤ 4 x ULN)

  * (Note: Patients with liver test abnormalities attributable to hepatic involvement by ALL will be permitted if the TBili is ≤ 5 x ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x institutional ULN

  * (Note: Patients with liver test abnormalities attributable to hepatic involvement by ALL will be permitted if the ALT/AST are ≤ 8 x ULN)
* Calculated creatinine clearance of > 30 ml/min/1.73m^2, as measured by the Modification of Diet in Renal Disease (MDRD) equation, will be eligible
* As patients with ALL frequently have cytopenias, no hematologic parameters will be required for enrollment or to receive the first cycle of treatment. However, adequate recovery of blood counts will be required to receive subsequent cycles
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2. (Performance status of 3 will be allowed if poor performance status is thought to be directly secondary to ALL)
* Ability to give informed consent and comply with the protocol
* Anticipated survival of at least 3 months, independent of ALL
* Female subjects of reproductive potential must agree to use an effective method of birth control from the time of signing the consent form until one of the following:

  * For subjects not expected to receive rituximab (i.e., CD20-negative): at least 3 weeks after the last dose of ponatinib, or
  * For subjects expected to receive rituximab (i.e., CD20-positive): at least 12 months after the last dose of rituximab
  * A subject does not have reproductive potential if they are (1) surgically sterilized, or (2) postmenopausal (i.e., a female who is > 50 years old or who has not had menses for ≥ 1 year), or (3) not heterosexually active
* Male subjects must agree to use an effective method of birth control and to not donate sperm from the time of signing the consent form until at least 3 weeks after the last dose of ponatinib

Exclusion Criteria:

* Burkitt lymphoma/leukemia
* No prior systemic therapy for ALL except to control acute symptoms and/or hyperleukocytosis (e.g., corticosteroids, cytarabine, etc.)
* No isolated extramedullary or known parenchymal central nervous system (CNS) disease
* History of acute pancreatitis within 1 year of enrollment or known chronic pancreatitis
* Symptomatic atherosclerotic cardiovascular disease (e.g., myocardial infarction, cerebrovascular accident, peripheral arterial disease, etc.) within 1 year of enrollment
* Active resistant hypertension, defined as having an ambulatory blood pressure above goal despite use of 3 antihypertensive medications from different classes
* Venous thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months of enrollment
* Known hypersensitivity or intolerance to any of the agents under investigation
* Other medical or psychiatric conditions that in the opinion of the investigator would preclude safe participation in the protocol
* May not be pregnant or nursing. Pregnancy test is only required in females, unless they do not have reproductive potential. For subjects not expected to receive rituximab (i.e., CD20-negative), nursing can occur 1 week after the last dose of ponatinib. For subjects expected to receive rituximab (i.e., CD20-positive), nursing can occur 6 months after the last dose of rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complete molecular response | Up to completion of 4 cycles (approximately 3 months) (cycle length = 21 days)
  Will be evaluated by BCR::ABL1 reverse transcriptase polymerase chain reaction.

SECONDARY OUTCOMES:
Incidence of non-hematologic toxicities greater than or equal to grade 3 | Up to 30 days after last dose of study treatment
  Will be graded in severity according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be reported as ratios/percentages. Will exclude asymptomatic grade 3 laboratory abnormalities.
Incidence of serious adverse events | Up to 30 days after last dose of study treatment
  Will be graded in severity using NCI CTCAE v 5.0. Will be reported as ratios/percentages.
Frequency of patients unable to complete one full cycle of etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin +/- rituximab + ponatinib (Feasibility) | Up to 5 years after last dose of study treatment
  Will be assessed descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present).
Event-free survival | Up to 5 years after last dose of study treatment
  Will be assessed descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present). Kaplan-Meier curves will be used to depict survival.
Relapse-free survival | Up to 5 years after last dose of study treatment
  Will be assessed descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present). Kaplan-Meier curves will be used to depict survival.
Duration of remission | Up to 5 years after last dose of study treatment
  Will be assessed descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present). Kaplan-Meier curves will be used to depict survival.
Overall survival | Up to 5 years after last dose of study treatment
  Will be assessed descriptively, using means and associated confidence intervals for continuous measures, simple ratios and Clopper-Pearson confidence intervals for binary measures, and either Kaplan-Meier or cumulative incidence estimates for time-to-event outcomes (depending on whether competing risks are present). Kaplan-Meier curves will be used to depict survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Cassaday, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No